CLINICAL TRIAL: NCT00505245
Title: Measuring the Symptom Distress of Cancer Patients: Development of a New Assessment System
Brief Title: New Assessment System in Measuring Symptom Distress in Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bayer (Industry); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry); Genentech, Inc. (Industry); Merck Sharp & Dohme LLC (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: BS99-094; NCI-2018-02461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BS99-094 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R01CA205146 (NIH)
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Caregiver; Health Care Provider; Malignant Neoplasm; Physician
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, QOL assessment, interview): Participants complete questionnaires and quality of life assessments, and may also complete interviews over 45 minutes periodically.
  Interventions: Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Complete interview
Other: Quality-of-Life Assessment — Complete quality of life assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies how well a new assessment system (MDASI or other MD Anderson-developed PRO instrument) works in measuring symptoms and the impact on quality of life in cancer patients. Development of a new assessment system may provide more information about the common symptoms that may occur in patients due to cancer and its treatment and how the symptoms impact quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine how the MD Anderson Inventory (MD Anderson Symptom Inventory [MDASI]) or other MD Anderson-developed patient reported outcome (PRO) instrument performs in various sample populations including community dwelling adults and patients who have different cancer types, who have undergone various treatments, and who have different and/or more severe symptoms.

II. To evaluate the MDASI or other MD Anderson-developed PRO instrument as an estimate of functional status and quality of life.

III. To assess the impact of symptom severity on standard function and health-related quality of life measures, including both quantitative and qualitative measures (patient interviews).

IV. To assess the pattern and severity of symptoms over multiple time points in order to assay the system's responsiveness to changes due to therapy or disease.

V. To explore the utility of an interactive voice response (IVR) system in enhancing the clinical care of outpatients.

VI. To explore the effect of information from an IVR symptom assessment system on the pattern of care and development of interdisciplinary protocols.

VII. To explore the feasibility of developing symptom management pathways for patients based on these symptom and quality of life data.

OUTLINE:

Participants complete questionnaires and quality of life assessments, and may also complete interviews over 45 minutes periodically.

ELIGIBILITY:
Inclusion Criteria:

* NORMAL SAMPLES: Community dwelling adults 18 years of age or older
* PATIENT SAMPLES: Inpatients and outpatients 18 years of age or older, being followed at UT MD Anderson
* EXPERT PANEL PROFESSIONAL PARTICIPANTS: Physician or other healthcare provider with at least 5 years of experience caring for patients with the disease and/or treatment of interest, at least one publication in the last 5 years dealing with the disease and/or treatment of interest (physician only), ability to speak and read English, consent to participate
* EXPERT PANEL FAMILY CAREGIVERS PARTICIPANTS: Identification as a family caregiver by patient enrolled as expert panel participant with the disease and/or treatment of interest, 18 years of age or older, ability to speak and read English, consent to participate
* EXPERT PANEL PATIENT PARTICIPANTS: Patient with identified family caregiver participating on Expert Panel, willingness to receive packet for expert panel participation

Exclusion Criteria:

* EXPERT PANEL PATIENT PARTICIPANTS: Patient with identified family caregiver participating on expert panel, willingness to receive packet for expert panel participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults, inpatients and outpatients with cancer being followed at University of Texas (UT) MD Anderson
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 1999-04-13 (Actual); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory (MDASI) tool or other MD Anderson-developed patient reported outcome (PRO) instrument validity | Up to 21 years
  Each item is rated 0 to 10 with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imaged or complete interference. The symptom severity and interference sub scales are mean values of the items in each scale. Hence the range of each sub scale is also 0 to 10. Lower values represent a better outcome. Higher values represent a worse outcome. The symptom severity and interference sub scales are not combined to compute a total score.
MD Anderson Symptom Inventory (MDASI) tool or other MD Anderson-developed PRO instrument reliability. | Up to 21 years
  Each item is rated 0 to 10 with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imaged or complete interference. The symptom severity and interference sub scales are mean values of the items in each scale. Hence the range of each sub scale is also 0 to 10. Lower values represent a better outcome. Higher values represent a worse outcome. The symptom severity and interference sub scales are not combined to compute a total score.
MD Anderson Symptom Inventory | Baseline up to 21 years
  Mean ratings of 11-point 0-10 scales; lower mean score = better outcome.
Eastern Cooperative Oncology Group Functional Status scale | Baseline up to 21 years
  6-point 0-5 scale; lower score = better outcome.
EuroQOL 5 Dimensions questionnaire | Baseline up to 21 years
  Scored on 5-point 1 to 5 scales; combined scores converted to index value for US = -0.573 to 1; higher values = better outcome.
The change in the symptom severity and interference with the function | Baseline up to 21 years
  Changes in patients' symptoms over time will be determined by differences in symptom severity scores on the MD Anderson Symptom Inventory MDASI collected at multiple time points. 0 to 10 with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imaged or complete interference. The symptom severity and interference sub scales are mean values of the items in each scale. Hence the range of each sub scale is also 0 to 10. Lower values represent a better outcome. Higher values represent a worse outcome. The symptom severity and interference sub scales are not combined to compute a total score.
MD Anderson Symptom Inventory (MDASI) tool or other MD Anderson-developed PRO instrument sensitivity | Up to 21 years
  Each item is rated 0 to 10 with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imaged or complete interference. The symptom severity and interference sub scales are mean values of the items in each scale. Hence the range of each sub scale is also 0 to 10. Lower values represent a better outcome. Higher values represent a worse outcome. The symptom severity and interference sub scales are not combined to compute a total score.
The quality of life questionnaire will be assessed. | Up to 21 years
  The European Organization for Cancer Treatment and Research Quality of Life scale (EORTC QLQ-C30) is a quality of life questionnaire that measures five functional areas (physical, social, role, cognitive, and emotional), eight symptoms (fatigue, nausea/vomiting, pain, dyspepsia, sleep disturbance, diarrhea, appetite loss, and constipation), financial impact, and overall quality of life. All of the sub scales and single-item measures range in score from 0 to 100 according to scoring algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org